With Love: Using Promotoras for a Hispanic Community Palliative Care Promotora Palliative Care

NCT03736031 March 28, 2019

## Statistical Analysis

- SAS 9.4 software (SAS Institute, Inc., Cary, North Carolina) was used to analyze the data.
- The average FACIT-Pal total scores were calculated for the promotora and the self-study groups at two points in time: before and after the intervention.
- Averages were reported along with standard deviations (SD).
- The average differences in FACIT-Pal total scores over time (after score minus before score) were calculated for the promotora and the standard of care groups and a two-sample independent *t*-test was performed. An alpha of 0.05 was used.